CLINICAL TRIAL: NCT04874779
Title: Risk of Acute Kidney Injury Among Patients Infected With COVID-19: A Retrospective Single Center Study
Brief Title: Acute Kidney Injury Risk in COVID-19
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Collaborators: University of Ha'il , Saudi Arabia. (Unknown)
Responsible Party: Principal Investigator, Mohamed E Ghoniem, Clinical Professor - Associate Professor of Internal Medicine- Faculty of Medicine, Zagazig University
Other Study IDs: COVID-1927
Record Dates: First submitted 2021-05-02; First posted 2021-05-06 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-05

CONDITIONS: Sever Acute Respiratory Syndrome and Acute Kidney Injury; Acute Kidney Injury
Keywords: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acute kidney injury (AKI) group: Acute kidney injury (AKI) group met the guidelines of Kidney Disease, Improving Global Outcomes (KDIGO)
  Interventions: Other: non
- NON-Acute kidney injury (non-AKI) group: NON-Acute kidney injury (non-AKI) group not met the guidelines of Kidney Disease Improving Global Outcomes (KDIGO)
  Interventions: Other: non

INTERVENTIONS:
Other: non — follow up investigations

SUMMARY:
Background. Within a year, COVID-19 has advanced from being an outbreak to a pandemic, spreading rapidly and globally with devastating impact. Currently, there is an ongoing debate among scientists about the pathophysiological relationship between COVID-19 and acute kidney injury (AKI). While a few studies have concluded that the mechanisms of AKI in COVID-19 patients are seemingly multifactorial and have not been fully explicated, others asserted that AKI remains rare among COVID-19-related diseases. Considering this knowledge-gap and its potential impact on the management of COVID-19-associated AKI, our study aims to explore the prevalence of AKI and to identify possible risk factors associated with AKI development among COVID-19 hospitalized patients. Materials and Methods. This retrospective cohort study included 83 patients with COVID-19 hospitalized at AL-AHRAR Hospital, Zagazig, Egypt, between June and August,2020. Exclusion criteria were: patients younger than 18 years of age; diagnosed with end stage kidney disease; placed on maintenance dialysis; booked for a kidney transplant or on nephrotoxic medications. All patients included in the study underwent complete blood count; liver and renal function tests; examination of hemostasis parameters; inflammatory markers; serum electrolytes; routine urinalysis; arterial blood gas and non-enhanced chest and abdominal computer tomography (CT) scans

DETAILED DESCRIPTION:
2.1. Study design and participants. Retrospective observational single-center study, including (83) laboratory-confirmed COVID-19 patients (age ≥ 18 years), hospitalized and isolated in the medical departments of AL-AHRAR Hospital, Zagazig, Egypt, from June 23 to August 29, 2020. All patients were isolated in the medical departments. None of them were admitted to the ICU or underwent mechanical ventilation. According to the WHO guidelines, a confirmed diagnosis of COVID-19 was defined as a positive result of a quantitative real-time reverse-transcriptase-polymerase chain reaction (RT-PCR) detection in a nasopharyngeal swab. (9) We excluded the following from this study: patients younger than 18 years, patients diagnosed with chronic kidney disease before admission, patients on maintenance dialysis or awaiting renal transplantation and patients taking any nephrotoxic medications a week prior to admission.

2.2. Data collection. The patients' medical history, underlying diseases, medications administered at home and in hospital, laboratory data, non-enhanced chest and abdominal computer tomography (CT) scans, were retrieved from electronic medical records. According to the Ministry of Health and Population (MOHP), Egypt Management protocol for COVID-19 Patients, version 1.4, 30th May,2020, (10), all patients received standard of care treatment including: (a) oxygen supply to achieve SaO2 ≥ 90%; (b) Hydroxychloroquine (400 mg twice in first day then 200 mg twice for 6 days); (C) Vitamin C (1gm daily); (d) Zinc (50mg daily); (e) Acetylcysteine 200 mg t.d.s.; (f) lactoferrin one sachet twice daily; (g) Anticoagulation if D-dimer > 1000.

2.3. Molecular detection of SARS-CoV-2 (RT-PCR). SARS-CoV-2 real-time reverse transcription polymerase chain reaction (RT-PCR) testing was performed on nasopharyngeal swabs using Thermofisher SCIENTIFIC's TaqPathTM COVID 19 CE IVD RT PCR Kit, 1000 reactions (Cat. No. A48067). The QUIAGEN extraction kit was used to extract viral RNA. Using Quick Dx Applied Biosystems 7500 real-time PCR instruments, the purified nucleic acid was reverse transcribed into cDNA and amplified using the TaqPathTM COVID 19 RT PCR Kit in one stage. Probes annealed to three unique SARS-CoV-2 target sequences: ORF1ab, nucleocapsid (N), and spike (S) primers/probes for bacteriophage MS2. The result was deemed null because two of the three genes and the MS2 (positive control) were all positive. COVID-19 was diagnosed whenever a positive real-time RT-PCR result was identified.

2.4. Laboratory procedures. Laboratory data included complete blood count by automated blood counter, liver and renal function tests by colorimetric method, examination of hemostasis parameters, inflammatory markers, serum Na, Serum K, serum Ca, urine dipstick test and arterial blood gas analysis.

2.5. Definitions. Acute kidney injury (AKI) was identified according to the guidelines of Kidney Disease Improving Global Outcomes (KDIGO). It is defined as any of the following: (I) an S.cr increase ≥0.3 mg/dL (≥26.5 μmol/L) within 48 h; or (II) an S.cr increase to ≥1.5 times baseline within the previous 7 days; or (III) a urine volume ≤0.5 mL/kg/h for 6 h. AKI is staged for severity according to the criteria presented in Table (1). (11) Urine output criteria were not used consistently for the diagnosis of AKI due to a lack of daily urine measurement in the electronic chart.

The Sequential Organ Failure Assessment (SOFA) score was developed as a morbidity severity score to focus on organ dysfunction, which can reliably predict disease severity and outcome. It includes 6 variables, each representing an organ system presented in Table (2). (12) Statistical Analyses. The SPSS software, version 26, was used for statistical analysis. ANOVA and univariate logistic regression analysis [odds ratio (OR) and 95% confidence intervals (CI)] were performed (significance level: P < 0.05).

Ethics statement. In order to maintain and ascertain the rights of patients without jeopardizing their privacy and confidentiality, informed verbal consents, in lieu of written informed consents, were obtained directly from all patients or their relatives. The requirements to obtain written informed consents were not attainable due to the inherent hazardous and contagious nature of COVID-19 epidemic, the strict restrictions by the hospital management, and the urgency of collecting the data.

ELIGIBILITY:
Inclusion Criteria:

According to the WHO guidelines, a confirmed diagnosis of COVID-19 was defined as a positive result of a quantitative real-time reverse-transcriptase-polymerase chain reaction (RT-PCR) detection in a nasopharyngeal swab.

Exclusion Criteria:

patients younger than 18 years, patients diagnosed with chronic kidney disease before admission, patients on maintenance dialysis or awaiting renal transplantation and patients taking any nephrotoxic medications a week prior to admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients' medical history, underlying diseases, medications administered at home and in hospital, laboratory data, non-enhanced chest and abdominal computer tomography (CT) scans, were retrieved from electronic medical records. According to the Ministry of Health and Population (MOHP), Egypt Management protocol for COVID-19 Patients, version 1.4, 30th May,2020, (10), all patients received standard of care treatment including: (a) oxygen supply to achieve SaO2 ≥ 90%; (b) Hydroxychloroquine (400 mg twice in first day then 200 mg twice for 6 days); (C) Vitamin C (1gm daily); (d) Zinc (50mg daily); (e) Acetylcysteine 200 mg t.d.s.; (f) lactoferrin one sachet twice daily; (g) Anticoagulation if D-dimer > 1000.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2020-11-18 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
The development of acute kidney injury or not following COVID-19 | 2 months after enrollement

CONTACTS AND LOCATIONS:
Overall Officials: mohamed ghonim, Principal Investigator — Associate professor of Internal Medicine , faculty of medicine, Zagazig University
Locations (1):
- Faculty of Medicine -Zagazig University, Zagazig, Egypt